CLINICAL TRIAL: NCT07221994
Title: The Effects of Blood Flow Restriction Combined With Low-Intensity Recumbent Stepping in Individuals With Advanced Parkinson's Disease
Brief Title: Blood Flow Restriction and Exercise in Parkinson's Disease
Acronym: BFR-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-44253
Record Dates: First submitted 2025-08-19; First posted 2025-10-29 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Parkinson' Disease
Keywords: Parkinson's disease; blood flow restriction; falls; postural instability; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Aerobic exercise (Nu-Step) recumbent stepping and blood flow restriction (BFR) (Experimental): Intervention (aerobic exercise + lower-extremity BFR)
  Interventions: Device: Blood flow restriction (BFR) and aerobic exercise via recumbent stepping (Nu-Step)

INTERVENTIONS:
Device: Blood flow restriction (BFR) and aerobic exercise via recumbent stepping (Nu-Step) — This intervention involves the combined application of training with BFR and aerobic exercise via recumbent stepping on a Nu-Step machine. The intervention will be administered to all study participants, twice-weekly, for 8 weeks.

SUMMARY:
The goal of this clinical trial is to learn whether training with blood flow restriction (BFR), combined with aerobic exercise (performing stepping on a Nu-Step exercise machine), can help improve mobility and other outcomes in people with progressed Parkinson's disease. The investigators hypothesize that training with BFR and aerobic exercise will produce enhanced outcomes related to mobility and quality of life.

BFR uses inflatable cuffs placed on participants' upper legs to gently reduce blood flow to the legs while exercising. This has been shown in studies in older adults and Parkinson's disease to improve strength while training with lighter loads, which may be helpful for people with Parkinson's.

Participants will be asked to complete 2 weekly training sessions (approximately 30 minutes each) for 8 weeks consisting of supervised aerobic stepping exercise on a Nu-step machine with BFR application during timed intervals. In addition to the training sessions, participants will be asked to periodically perform confidential surveys and tests related to function and disease symptoms, and wear a provided smartwatch (which can be kept upon successful completion of the study). All sessions involve individual monitoring and medical supervision by licensed physical therapists as well as access to all necessary equipment.

DETAILED DESCRIPTION:
This study's primary objective is to determine the exploratory safety of the combined recumbent stepping + BFR intervention for this population. Secondary aims are to evaluate the exploratory efficacy on the intervention for Parkinson's symptoms including functional mobility, autonomic function, daily step counts, cognition, and quality of life, as well as obtain feasibility and acceptability of the intervention from participants.

This is a pilot clinical trial (pre-post) which will investigate the safety, feasibility, and exploratory effectiveness of a novel, 8-week clinical trial with BFR + low-intensity recumbent stepping for advanced PD in 4 participants. Data will be collected at three time-points: baseline, after the 8-week intervention, and at 4-weeks post-intervention cessation to assess for continued longitudinal intervention effects and short-term durability. Findings will guide optimization, scalability, and future clinical implementation via larger randomized controlled trials and protocol refinement as appropriate.

Screening, consent, and baseline assessments will be conducted individually with the PI; all participants will continue their prescribed Parkinson's medications during the study. Participants will be given a fitness tracker watch and training as needed, then complete the 8-week intervention with continuous monitoring by one of the investigators using heart rate, SpO2, rate of perceived exertion (RPE), and blood pressure (BP) taken before and/or during and after the intervention.

BFR Intervention Details: Participants will perform recumbent stepping (legs only) using a Nu-Step machine as detailed above, with Fit Cuffs®' BFR straps wrapped around their bilateral proximal thighs at 40% arterial occlusion pressure (remaining consistent throughout the protocol). The arterial occlusion pressure at rest (rAOP) will be assessed using a FitCuffs® pressure system and pulse oximeter. The cuffs will be inflated until the distal pulse (measured at the toe) is no longer detectable. The corresponding pressure will be recorded as the rAOP and used to calculate the BFR training pressure at 40% rAOP. In the case of issue using the device, a doppler ultrasound will be used at the dorsalis pedis artery to check for occlusion and associated pressure.

Weekly surveys will be emailed to participants for input of their daily (averaged) step counts during that week, falls, heart rate variability, and feedback regarding the intervention, with participant follow-up performed by the investigators as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. People with advanced Parkinson's disease. "Advanced PD" will include signs of progressed disease including orthostatic hypotension and/or motor issues reflective of postural instability and/or mild-moderate bilateral symptoms (confirmed visually in clinic or home by a medical provider such as an MD/PT and/or documented in the medical record.
3. Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
4. Diagnosis of idiopathic Parkinson's disease (self-reported okay, documented preferred)
5. Independent ambulation (≥10m with or without an assistive device)
6. Commitment to participate in the exercise intervention as outlined
7. Score of ≥21 on the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

1. History of cardiovascular disease, uncontrolled hypertension (blood pressure

   ≥140/90 mmHg), deep-vein thrombosis, varicose veins, or rhabdomyolysis which a patient's primary physician determines would preclude them from safe study participation.
2. Ankle branchial index ≤ 0.9 or > 1.3
3. History of or comorbid conditions spanning cardiovascular, neurological, or orthopedic injuries which may prevent for the safe administration of the intervention (a healthcare provider's clearance or guidance will be obtained in these situations to ensure appropriateness), including current medications.
4. History of uncontrolled diabetes, BMI > 40, or severe cognitive impairment (as measured by MoCA <21)
5. Atypical PD diagnoses or ON PD-medication worsening of motor symptoms
6. Absolute contraindications to exercise as per the American College of Sports Medicine (uncontrolled arrhythmias, third-degree heart block, recent electrocardiogram (EKG) changes, unstable angina, acute myocardial infarction, or acute congestive heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by Custom Survey & Vitals Monitoring during & post-intervention | Participants will be monitored continuously during each session (vitals and response via subjective report), then each week, throughout the 8-week study intervention and 4-weeks post-intervention.
  Treatment-Related Adverse Events will be assessed during session using heart rate (HR), rate of perceived exertion (RPE), and subjective interview for tolerance, fatigue, and pain, as well as use a Custom Qualtrics survey which each participant will fill out each week to illuminate potential adverse events and whether they had worsening of PD motor symptoms, changes in sleep or activity scores, and/or something they would like to disclose to study personnel (free text reponse).

SECONDARY OUTCOMES:
Overall PD motor severity | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  The Unified Parkinson's Disease Rating Scale Motor subscore (UPDRS-III) will be used to determine changes in individuals' overall PD motor severity.
Improvement of functional mobility | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  The "Timed up and Go" test (TUG); single and dual-tasking components will be used to determine whether changes are observed in functional mobility.
Improvement of functional mobility | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  The 5x sit to stand test will be used to assess for changes in functional mobility.
Improvement of fall incidence | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  The number of falls averaged and self-reported by the patient each week will be captured at baseline, then captured throughout the intervention and post-intervention observation period using custom Qualtrics survery which inquires about falls per week.
Improvement of orthostatic incidence | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  The number of episodes of orthostatic hypotension averaged and self-reported by the patient each week will be captured at baseline, then captured throughout the intervention and post-intervention observation period using custom Qualtrics survery which inquires about orthostatic hypotension per week.
Improvement of daily activity (step) counts | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  The number of daily steps averaged and self-reported using the provided study wearable by the patient each week will be captured at baseline, then throughout the intervention and post-intervention observation period using a custom Qualtrics survery which asks participants to self-report (using the smartwatch) averaged step counts.
Improvement of cognition | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  Participant cognition will be measured using the MoCA exam (Montreal Cognitive Exam).
Improvement of cognition | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  Participant cognition will be measured using the Trail-Making-Test (TMT) either online or in-person by the trained PIs.
Improvement of Parkinson's disease related quality of life | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  Participant cognition will be measured using the PD-specific quality of life (PDQ-8) self-reported clinical metric
Improvement of lower-extremity muscle strength | Baseline, 8 weeks following intervention start, then 4 weeks after the end of the intervention (12 weeks total following intervention start).
  Participant strength will be measured using dynamometer testing of quadriceps and hamstrings muscles
Intervention Adherence | 12 weeks total following intervention start-last study data collection point; throughout during 8-week intervention (weekly) using custom Qualtrics Survey.
  This will be assessed using PI/participant tracking of the amount of protocol sessions attended by participants.
Participant experience of the intervention | 12 weeks total following intervention start-last study data collection point; throughout during 8-week intervention (weekly) using custom Qualtrics Survey.
  Participant experience and perceptions with the intervention will be assessed formally with participant feedback using the summative custom Qualtrics survey via open-ended feedback at the end of the study, as well as informally throughout the study during live conversations with the PIs.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Bath, DPT, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Health & Wellness Center (UCSF Mission Bay), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated participant data which has been de-identified; likely provided through descriptive statistics and aggregated results only, due to the relatively small sample size to prevent potential identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months following study completion.
Access Criteria: Researchers and other interested parties will be asked to contact the PI via email. Data will only be shared as detailed above (aggregated, de-identified data) in alignment with UCSF IRB protocol.

REFERENCES:
- [Background] Chang HC, Lu CS, Chiou WD, Chen CC, Weng YH, Chang YJ. An 8-Week Low-Intensity Progressive Cycling Training Improves Motor Functions in Patients with Early-Stage Parkinson's Disease. J Clin Neurol. 2018 Apr;14(2):225-233. doi: 10.3988/jcn.2018.14.2.225. PMID 29629527
- [Background] Liao JY, Bohnen NI. Is heart rate variability the heart of the matter for freezing of gait? Parkinsonism Relat Disord. 2023 Aug;113:105763. doi: 10.1016/j.parkreldis.2023.105763. Epub 2023 Jul 11. No abstract available. PMID 37468360
- [Background] Chen Z, Li G, Liu J. Autonomic dysfunction in Parkinson's disease: Implications for pathophysiology, diagnosis, and treatment. Neurobiol Dis. 2020 Feb;134:104700. doi: 10.1016/j.nbd.2019.104700. Epub 2019 Dec 3. PMID 31809788
- [Background] Douris PC, Cogen ZS, Fields HT, Greco LC, Hasley MR, Machado CM, Romagnuolo PM, Stamboulis G, DiFrancisco-Donoghue J. THE EFFECTS OF BLOOD FLOW RESTRICTION TRAINING ON FUNCTIONAL IMPROVEMENTS IN AN ACTIVE SINGLE SUBJECT WITH PARKINSON DISEASE. Int J Sports Phys Ther. 2018 Apr;13(2):247-254. PMID 30090683
- [Background] Manago MM, Cohen ET, Alvarez E, Hager ER, Owens JG, Bade M. Feasibility of Low-Load Resistance Training Using Blood Flow Restriction for People With Advanced Multiple Sclerosis: A Prospective Cohort Study. Phys Ther. 2024 Jan 1;104(1):pzad135. doi: 10.1093/ptj/pzad135. PMID 37815934
- [Background] Lopes KG, Farinatti P, Bottino DA, DE Souza MDGC, Maranhao PA, Bouskela E, Lourenco RA, DE Oliveira RB. Does Resistance Training with Blood Flow Restriction Affect Blood Pressure and Cardiac Autonomic Modulation in Older Adults? Int J Exerc Sci. 2021 Apr 1;14(3):410-422. doi: 10.70252/OXXF4710. eCollection 2021. PMID 34055161
- [Background] Franz A, Ji S, Bittersohl B, Zilkens C, Behringer M. Impact of a Six-Week Prehabilitation With Blood-Flow Restriction Training on Pre- and Postoperative Skeletal Muscle Mass and Strength in Patients Receiving Primary Total Knee Arthroplasty. Front Physiol. 2022 Jun 14;13:881484. doi: 10.3389/fphys.2022.881484. eCollection 2022. PMID 35774280